CLINICAL TRIAL: NCT05459805
Title: Multicenter Clinical Study on the Optimal Treatment Protocol and Outcome of Cough Variant Asthma With Chinese and Western Medicine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Collaborators: Xin Hua Hospital of Zhejiang Province (Other); Hangzhou Hospital of Traditional Chinese Medicine (Other); Affiliated Wenling Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022ZZ011; ChiCTR2100048636 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2022-07-06; First posted 2022-07-15 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2022-07

CONDITIONS: Cough Variant Asthma
Keywords: cough variant asthma; traditional Chinese medicine; clinical trial
MeSH Terms: conditions — Cough-Variant Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): those receive ICS/LABA plus traditional Chinese medicine
  Interventions: Drug: traditional chinese medicine Xuanfei-Zhike formula; Drug: inhaled corticosteroids (ICS) and long-acting β2-agonist (LABA)
- group 2 (Active Comparator): those receive ICS/LABA alone
  Interventions: Drug: inhaled corticosteroids (ICS) and long-acting β2-agonist (LABA)

INTERVENTIONS:
Drug: traditional chinese medicine Xuanfei-Zhike formula — 200ml, bid, for 8 weeks
  Arms: group 1
Drug: inhaled corticosteroids (ICS) and long-acting β2-agonist (LABA) — one suction, q12h, for 8 weeks

SUMMARY:
To explore the disease outcome prognosis of cough variant asthma by observing the outcomes of cough variant asthma and the effects of Chinese and Western medicine interventions, and to provide a scientific basis for optimizing the treatment protocol of combined traditional and Western medicine for cough variant asthma. This is a multi-center, non-randomized, prospective cohort study. This study started in March 2022 and is going on now. On an informed consent basis, a cohort of 164 patients with diagnosis of CVA are engaged. All patients will receive 8-week treatment (ICS/LABA plus Chinese herbal medicine for trial group while ICS/LABA only for control group) and be observed in next 24 weeks. Patients will be followed up every 2 weeks during treatment period and every 4 weeks in observation.The feasibility and correctness of the study will be supervised by two supervisors. To ensure that participants adhere to their follow-up plans, we remind them of their fixed visiting by phone or message. Additionally, incentives are used to appreciate participants for their cooperation.

ELIGIBILITY:
Inclusion Criteria:

1. conform to diagnosis of CVA;
2. 18 years≤age≤65 years;
3. agree to participant in this trial.

Exclusion Criteria:

1. comorbidity of respiratory and pulmonary infections;
2. history of mental illness;
3. comorbidity of heart and cardiovascular, liver, kidney and hematopoietic function and other severe diseases;
4. participants of other clinical trials who may make a difference in our trial;
5. treatment with other Chinese herb.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
total effective rate calculated by the Cough-related Symptom Scale | week 8
  Cough-related Symptom Scale is specially designed for this trial. Question1-5 in CSS comes from Chinese national guideline on diagnosis and management of cough (2021) and the rest questions are set based on clinical experience and other study . Total effective rate can be directly reflected in Efficacy Index (EI) which set by National Medical Products Administration .
total effective rate calculated by the Cough-related Symptom Scale | week 32
  Cough-related Symptom Scale is specially designed for this trial. Question1-5 in CSS comes from Chinese national guideline on diagnosis and management of cough (2021) and the rest questions are set based on clinical experience and other study . Total effective rate can be directly reflected in Efficacy Index (EI) which set by National Medical Products Administration .

SECONDARY OUTCOMES:
change from baseline in Cough-related Symptom Scale | baseline and week 8 ,baseline and week 32
  This scale consists of two parts. Question1-5 come from Chinese national guideline on diagnosis and management of cough (2021) to evaluate the symptom of cough. Question6-10 are some accompanying performances, including cough-stimulated factors like wind, cold air, smoking etc, sputum, sensations of "persistent tickling", "thirsty", "Qi inversion" in throat.
change from baseline in Cough severity visual analogue scale | baseline and week 8 ,baseline and week 32
  Cough severity visual analogue scale (VAS) is used to record participants' assessments of cough severity. It is shown as a 0-mm to 100-mm liner scale ranging from "no cough" to "severe cough". The bigger score represents more severe cough.
change from baseline in Leicester Cough Questionnaire | baseline and week 8 ,baseline and week 32
  Leicester Cough Questionnaire, as a useful tool in clinical trial, consists of 19 items which is a repeatable, valid self-evaluated quality of life measure of chronic cough and responsive to change .
change from baseline in Pulmonary function | baseline and week 8 ,baseline and week 32
  Pulmonary function test reveals some details of a patient's condition in respiratory function, like forced vital capacity (FVC), forced expiratory volume in one second (FEV1), FEV1/FVC, peak expiratory flow (PEF), forced expiratory flow 25% (FEF25), forced expiratory flow 75% (FEF75), forced expiratory flow between 25% and 75% of forced vital capacity (FEF(25-75)) etc.
CVA recurrence rate from week 8 to week 32 | week 32
  CVA recurrence rate is defined as the occurance rate of similar cough which conforms to CVA diagnosis criteria during 6-month observation.
the ratio of progressing to typical asthma from week 8 to week 32 | week 32
  the ratio of progressing to typical asthma is characterized as the ratio of participants who turning from CVA into classic asthma based on Guidelines for bronchial asthma prevent and management (2020 edition) during 6-month observation.
change from baseline in fractional exhaled nitric oxide | baseline and week 8 ,baseline and week 32
  Nitric oxide (NO) is produced by inducible nitric oxide synthase (iNOS) in airway epithelial cells and FENO is associated with eosinophilic airway inflammation which usually indicates the sensitivity to ICS.
change from baseline in Serum IgE | baseline and week 8 ,baseline and week 32
  IgE is linked to its ability to affect several immune and structural cells involved in allergic asthma.

CONTACTS AND LOCATIONS:
Overall Officials: Junchao Yang, Study Chair — The First Affiliated Hospital of Zhejiang Chinese Medical University
Locations (4):
- China (4):
  - Hangzhou Hospital of Traditional Chinese Medicine, Hangzhou
  - The First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou
  - Xin Hua Hospital of Zhejiang Province, Hangzhou
  - The First People's Hospital of Wenling, Taizhou

IPD SHARING:
Plan to Share IPD: Yes
ndividual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. For individual participant data meta-analysis. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our Hospital's data warehouse but without investigator support other than deposited metadata.